CLINICAL TRIAL: NCT00138840
Title: A Randomized, Double-Blind, Placebo-Controlled Clinical Study of the Oral IL-12/23 Inhibitor, STA-5326 Mesylate, for the Induction of Clinical Response in Patients With Crohn's Disease
Brief Title: Study of STA-5326 Mesylate in Patients With Moderate to Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synta Pharmaceuticals Corp. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5326-07
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2008-12-04 (Estimated); Status verified 2008-12

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; Gastroenterology
MeSH Terms: conditions — Crohn Disease | interventions — apilimod

INTERVENTIONS:
Drug: STA-5326 mesylate

SUMMARY:
STA-5326 is an experimental drug that has been shown to block the release of interleukin-12 from peripheral blood mononuclear cells. Given this activity on the immune system, STA-5326 mesylate is a potential treatment for various autoimmune diseases, such as Crohn's disease, that are mediated by the inappropriate expression of Th1 cytokines.

This study is evaluating the use of STA-5326 mesylate in patients with moderate to severe, active Crohn's disease. Study visits include a screening visit, 9 treatment period visits over 6 months and a follow-up visit that will occur 30 days following the end of treatment. Study drug treatment will continue for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Is male or female aged 18 through 75 years.
* Has Crohn's disease diagnosed definitively prior to Screening (based upon clinical, endoscopic, radiologic imaging, or histological assessments).
* Has a Crohn's Disease Activity Index (CDAI) score of 220 to 450, inclusive at Baseline.

Exclusion Criteria:

* Has any clinically significant disease (eg, renal, hepatic, neurological, cardiovascular, pulmonary, endocrinologic, psychiatric, hematologic, urologic, or other acute or chronic illness) that, in the opinion of the investigator, would make the patient an unsuitable candidate for this study.
* Is a woman who has a positive pregnancy test, who is breast-feeding, or who is sexually active without using birth control during the course of the study and Follow-Up period.
* Is a woman of childbearing potential or a man who does not agree to use 2 forms of contraception during the course of the study and Follow-Up period.
* Has clinically significant hematologic, hepatic or renal laboratory abnormalities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282
Dates: Start 2005-08

PRIMARY OUTCOMES:
Proportion of patients achieving clinical remission and clinical response at Day 29

SECONDARY OUTCOMES:
Proportion of patients achieving: a clinical remission at Days 29 and 43
a clinical response from Baseline to Day 29 and from Baseline to Day 43
a reduction in endoscopic scores from Baseline to Day 29
an increase in the Inflammatory Bowel Disease Questionnaire (IBDQ) score from Baseline to Days 29 and 43
a clinical remission or clinical response at Days 29 and 43 in the subset of patients with elevated C-reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Sands, MD — Massachusetts General Hospital
Locations (35):
- United States (31):
  - Gastroenterology Associates, Little Rock, Arkansas
  - Advanced Clinical Research Institute, Anaheim, California
  - Community Clinical Trials, Orange, California
  - Medical Associates Research Group, San Diego, California
  - Southern Clinical Research Consultants, Hollywood, Florida
  - Borland Groover Clinic, Jacksonville, Florida
  - Miami Research Associates, Miami, Florida
  - Advanced Gastroenterology Highland Lakes Medical Center, Palm Harbor, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology, Atlanta, Georgia
  - Univ. of Louisville Clinical Research Unit, Louisville, Kentucky
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Capital Gastroenterology Consultants, P.A., Silver Spring, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Gastroenterology Research Associates, Cedar Knolls, New Jersey
  - Asher Kornbluth, MD, New York, New York
  - Rochester Institute for Digestive Diseases and Sciences, Inc., Rochester, New York
  - Asheville Gastroenterology Associates, PA, Asheville, North Carolina
  - Carolina Digestive Health Associates, Charlotte, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Wake Research Associates, LLC., Raleigh, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Columbia Gastroenterology Associates, P.A., Columbia, South Carolina
  - Gastroenterology Center of the MidSouth, Germantown, Tennessee
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Austin Gastroenterology, Austin, Texas
  - New River Valley Research Institute, Christiansburg, Virginia
  - Wisconsin Center for Advanced Research, Milwaukee, Wisconsin
- Canada (4):
  - University of Calgary Health Sciences, Calgary, Alberta
  - London Health Science Center South Street Campus, London, Ontario
  - London Health Science Center University Campus, London, Ontario
  - Saskatoon Medical Specialists, Saskatoon, Saskatchewan